CLINICAL TRIAL: NCT04457557
Title: Evaluation of the Effect of Local Anesthetic Concentration on Rebound Pain After Interscalene Block for Shoulder Surgery
Brief Title: Local Anesthetic Concentration and Rebound Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, In-kyong Yi, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MED-INT-20-140
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Rebound Pain
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial One group received interscalene block with 0.15% of ropivacaine One group received interscalene block with 0.5% of ropivacaine
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Only investigator who prepared the local anesthetics knows the group. Nerve block performer and outcome assessor are applied masking.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low concentration (Experimental): Interscalene block with 0.15% ropivacaine 15 ml
  Interventions: Other: Reduced concentration of local anesthetic (ropivacaine)
- Usual concentration (Active Comparator): Interscalene block with 0.5% ropivacaine 15 ml
  Interventions: Other: Usual concentration of local anesthetic (ropivacaine)

INTERVENTIONS:
Other: Reduced concentration of local anesthetic (ropivacaine) — Reduced concentration of ropivacaine We usually use 0.5% ropivacaine in our facility. The intervention group used 0.15% ropivacaine 15 ml
  Arms: Low concentration
Other: Usual concentration of local anesthetic (ropivacaine) — 0.5% ropivacaine 15ml
  Arms: Usual concentration

SUMMARY:
The rebound pain after nerve block could interfere with patient's recovery and rehabilitation. It is not known how local anesthetic concentrations affect rebound pain. The aim of this study is evaluation of the effect of local anesthetic concentration on rebound pain after interscalene block for shoulder surgery.

DETAILED DESCRIPTION:
Shoulder surgery is related to more than moderate pain after surgery. Interscalene nerve block could reduce the postoperative pain effectively. When the effect of nerve block ends, however, rebound pain could appear. The rebound pain could interfere with patient's recovery and rehabilitation.

The mechanism of rebound pain is not well known. One of possible mechanism is that the pain stimulus that was blocked suddenly comes out, and it is perceived as more severe pain. The strength of the block may vary depending on the concentration of the local anesthetic. Therefore, the concentration of local anesthetics could affect rebound pain. The aim of this study is evaluation of the effect of local anesthetic concentration on rebound pain after interscalene block for shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective shoulder surgery under general anesthesia and interscalene block for postoperative pain

Exclusion Criteria:

* Contraindication of interscalene block: pulmonary disease, lung resection history, brachial nerve injury
* Diabetic neuropathy
* Adverse drug reaction history to ropivacaine, fentanyl
* Impaired coagulation

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Rebound pain score | 48 hours after surgery
  It is calculated by subtracting the visual analogue scale (VAS) of pain at the last time when the nerve block was effective from the highest VAS for 12 hours from the time when the nerve block effect disappeared.
  VAS of pain: 0=no pain ~ 10=very severe pain

SECONDARY OUTCOMES:
total postoperative fentanyl dose | 48 hours after surgery
  Total dose of fentanyl injected (mcg) through patient controlled analgesia (PCA) for 48 hours after surgery
fentanyl bolus injection time | 48 hours after surgery
  Number of bolus injection times using patient controlled analgesia (PCA)
Subjective satisfaction | 48 hours after surgery
  Patient's subjective satisfaction 48 hours after surgery Use visual analogue scale (0=very unsatisfied, 10= very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: In Kyong Yi, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou university school of medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
We will provide it when we have a reasonable request.